CLINICAL TRIAL: NCT00564980
Title: A Randomized Prospective Study Comparing TFCC Debridement and Wafer Procedure With TFCC Debridement and Ulnar Shortening Osteotomy for Ulno-Carpal Abutment Syndrome. (UAS Study)
Brief Title: PRCT: Comparing Two Procedures for Ulno-Carpal Abutment Syndrome.
Acronym: UAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit required number of subjects.
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-061
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Joint Disease
Keywords: Randomized; Prospective; Procedure / Surgery
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Wafer Procedure
  Interventions: Procedure: Wafer Procedure
- 2 (Active Comparator): Ulnar shortening osteotomy
  Interventions: Procedure: Ulnar shortening osteotomy

INTERVENTIONS:
Procedure: Wafer Procedure — A dorsal approach to the distal ulna is used dividing the extensor retinaculum between the 5th and 6th compartments. The ulnar head is exposed through a transverse capsulotomy. Cartilage and bone are resected to result in slight negative ulnar variance based on the preoperative pronated grip view. The ulnar styloid and TFCC attachments are preserved. The dorsal capsule and retinaculum are repaired in separate layers.
  Arms: 1
Procedure: Ulnar shortening osteotomy — A longitudinal incision of approximately 8 cm is made at the distal third of the ulna along the ulnar border of the forearm. The interval between the flexor carpi ulnaris is used. The ulna is exposed at its distal third preserving the periosteum. Care is taken to protect the sensory branches of the lunar nerve. An oblique osteotomy is performed using a reciprocating saw, removing enough bone to result is slight negative ulnar variance. Fixation and compression at the osteotomy site is achieved using a 5 or 6 hole titanium LC-DCP plate.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate two different currently accepted surgical treatments for UAS (ulnocarpal abutment syndrome).

The hypothesis is that ulnar shortening osteotomy procedure will be associated with longer surgical time and increased complication rate when compared to the wafer procedure. It is unclear as to whether there will be a difference in functional outcome between the two groups.

DETAILED DESCRIPTION:
Ulnocarpal abutment syndrome (UAS) (also known as ulnar impaction syndrome, ulnocarpal impingement,ulnar carpal loading) is a common cause of ulnar sided wrist pain.

UAS results from increased loading of the ulnocarpal articulation and is usually associated with a positive ulnar variance. The increased loading of the joint can lead to degeneration and perforation of the Triangular fibrocartilage (TFC). Chondromalacic changes develop on the opposing surfaces of the lunate and triquetrum distally and the ulnar head proximally. A disruption of the lunotriquetral ligament may following with ensuing LT arthritis.

Treatment of UAS involves decompression of the pressure and impingement, or abutment of the ulnocarpal articulation. Debridement of triangular fibrocartilage complex (TFCC) tears alone in the patient with UAS may have a failure rate of as much as 25% to 30%. Good results have been reported with combined arthroscopic TFCC debridement and distal ulnar resection. 69% excellent and 32% good results have been reported with an open limited distal ulnar resection in patients with a TFCC tear and positive ulnar variance. Similar results have been reported with both ulnar shortening osteotomy and open wafer distal ulnar resections in the UAS patient. Because these treatment choices appear to yield similar relief of symptoms, determination of the optimal treatment protocol remains a point of debate.

The literature contains retrospective data comparing open wafer procedure with ulnar shortening osteotomies for the treatment of UAS. Likewise, the literature comparing arthroscopic wafer and ulnar shortening osteotomy is retrospective. However, there are, to date, no randomized prospective clinical trials comparing these types of surgery. Both types of surgery are widely accepted and the optimal treatment remains under debate. It is unclear how the techniques compare in terms of efficacy of elimination of symptoms of UAS and also in terms of relative complication rate.

ELIGIBILITY:
Inclusion Criteria:

* persistent ulnar-sided wrist pain of a minimum of 6 months duration despite conservative management
* a positive ulnocarpal stress test
* neutral or positive ulnar variance as measured from a standard posteroanterior radiograph of the wrist
* central TFCC perforation or lunate chondral damage consistent with UAS based on arthroscopic evaluation
* arthroscopically debrided TFCC tear

Exclusion Criteria:

* absence of a TFCC tear or lunate chondral damage
* repairable TFCC tear
* severe ulnocarpal arthrosis
* pre-operative diagnosis of clinically symptomatic scapholunate ligament (SL), lunotriquetral ligament (LT), or distal radioulnar joint (DRUJ) instability
* previous forearm or wrist fracture
* history of inflammatory arthritis
* presence of other wrist pathology
* a requirement for concomitant surgery for an unrelated condition
* skeletal maturity

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) at baseline, 6 weeks, 3, 6 and 12 months post-operatively. | Subjects are followed for 12 months post-op.

SECONDARY OUTCOMES:
Wrist range of motion, grip strength, radiographs and pain Visual Analog Scale | Baseline, 6 weeks, 3,6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand H Perey, MD, Principal Investigator — Royal Columbian Hospital, Eagle Ridge Hospital
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia

REFERENCES:
- [Background] Palmer AK, Glisson RR, Werner FW. Ulnar variance determination. J Hand Surg Am. 1982 Jul;7(4):376-9. doi: 10.1016/s0363-5023(82)80147-0. No abstract available. PMID 7119397
- [Background] Friedman SL, Palmer AK. The ulnar impaction syndrome. Hand Clin. 1991 May;7(2):295-310. PMID 1880164
- [Background] Tomaino MM. The importance of the pronated grip x-ray view in evaluating ulnar variance. J Hand Surg Am. 2000 Mar;25(2):352-7. doi: 10.1053/jhsu.2000.jhsu25a0352. PMID 10722828
- [Background] Hulsizer D, Weiss AP, Akelman E. Ulna-shortening osteotomy after failed arthroscopic debridement of the triangular fibrocartilage complex. J Hand Surg Am. 1997 Jul;22(4):694-8. doi: 10.1016/S0363-5023(97)80130-X. PMID 9260628
- [Background] Minami A, Kato H. Ulnar shortening for triangular fibrocartilage complex tears associated with ulnar positive variance. J Hand Surg Am. 1998 Sep;23(5):904-8. doi: 10.1016/S0363-5023(98)80171-8. PMID 9763270
- [Background] Feldon P, Terrono AL, Belsky MR. Wafer distal ulna resection for triangular fibrocartilage tears and/or ulna impaction syndrome. J Hand Surg Am. 1992 Jul;17(4):731-7. doi: 10.1016/0363-5023(92)90325-j. PMID 1629557
- [Background] Tomaino MM, Weiser RW. Combined arthroscopic TFCC debridement and wafer resection of the distal ulna in wrists with triangular fibrocartilage complex tears and positive ulnar variance. J Hand Surg Am. 2001 Nov;26(6):1047-52. doi: 10.1053/jhsu.2001.28757. PMID 11721249
- [Background] Constantine KJ, Tomaino MM, Herndon JH, Sotereanos DG. Comparison of ulnar shortening osteotomy and the wafer resection procedure as treatment for ulnar impaction syndrome. J Hand Surg Am. 2000 Jan;25(1):55-60. doi: 10.1053/jhsu.2000.jhsu025a0055. PMID 10642473
- [Background] Bernstein MA, Nagle DJ, Martinez A, Stogin JM Jr, Wiedrich TA. A comparison of combined arthroscopic triangular fibrocartilage complex debridement and arthroscopic wafer distal ulna resection versus arthroscopic triangular fibrocartilage complex debridement and ulnar shortening osteotomy for ulnocarpal abutment syndrome. Arthroscopy. 2004 Apr;20(4):392-401. doi: 10.1016/j.arthro.2004.01.013. PMID 15067279
- [Background] Milch H. Cuff resection of the ulna for malunited colles' fracture. JBJS (AM): 1941;23:311-313